CLINICAL TRIAL: NCT01524887
Title: A Phase 3 Randomized, Double-blind, Placebo-Controlled Study of the Safety and Effectiveness of Immune Globulin Intravenous (Human), 10% Solution (IGIV, 10%) for the Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Phase 3 IGIV, 10% in Alzheimer´s Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because the first Phase 3 did not demonstrate efficacy on the co-primary endpoints. The known safety profile remained unchanged.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161003; 2011-000914-21 (EudraCT Number)
Record Dates: First submitted 2012-01-20; First posted 2012-02-02 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer´s Disease
MeSH Terms: interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IGIV, 10% at high dose (0.4 g/kg) (Experimental)
  Interventions: Biological: Immune Globulin Intravenous (Human), 10% Solution
- IGIV, 10% at low dose (0.2 g/kg) (Experimental)
  Interventions: Biological: Immune Globulin Intravenous (Human), 10% Solution
- Placebo control (Placebo Comparator)
  Interventions: Biological: Human albumin 0.25%

INTERVENTIONS:
Biological: Immune Globulin Intravenous (Human), 10% Solution — Intravenous infusion every 2 weeks over 18 months
  Other Names: IGIV, 10%
  Arms: IGIV, 10% at high dose (0.4 g/kg); IGIV, 10% at low dose (0.2 g/kg)
Biological: Human albumin 0.25% — Intravenous infusion every 2 weeks over 18 months
  Arms: Placebo control

SUMMARY:
The purpose of this study is to provide evidence of efficacy and safety to support the development of IGIV, 10% as a treatment option for patients with mild to moderate Alzheimer´s Disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of age 50 to 89 years inclusive at the time of screening
* Written informed consent obtained from either the subject or the subject's legally authorized representative prior to any study-related procedures
* Written informed consent obtained from an able and competent caregiver who is willing to comply with the requirements of the protocol pertaining to him/her, including facilitating the subject's participation in the study
* Diagnosis of Probable Alzheimer´s Disease (AD) according to NINCDS-ADRDA* 1984 criteria (* National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association)
* Dementia of mild to moderate severity (Mini-Mental State Examination [MMSE] 16-26 inclusive at the time of screening)
* Neuroimaging (computed tomography [CT] or MRI) performed after symptom onset consistent with AD diagnosis
* Willingness to comply with the requirements of the protocol and ability to comply with testing and infusion regimen, including adequate corrected visual acuity and hearing ability
* For at least 12 weeks prior to screening, on stable doses of AD medication(s) approved by local regulatory authorities. Subjects must not be on two acetylcholinesterase inhibitors concurrently.
* Venous access for repeated infusion and phlebotomy
* If receiving psychoactive medications (eg, antidepressants other than monoamine oxidase inhibitors [MAOIs] and most tricyclics, antipsychotics, anxiolytics, anticonvulsants, mood stabilizers, etc.), must be on stable doses for at least 6 weeks prior to screening
* For women of childbearing potential, the subject must have a negative pregnancy test at screening and must agree to employ adequate contraceptive measures (eg, birth control pills/patches, intrauterine device, or diaphragm or condom [for male partner] with spermicidal jelly or foam) throughout the course of the study
* For subjects with a coronary artery stent, the subject must receive documented medical clearance from an interventional cardiologist stating that the subject is not at increased risk for stent occlusion with immunoglobulin treatment
* For subjects with an endovascular stent, the subject must receive documented medical clearance from a vascular surgeon stating that the subject is not at increased risk for thromboembolic events with immunoglobulin treatment

Main Exclusion Criteria:

* Possible AD by NINCDS-ADRDA criteria or non-Alzheimer dementia (eg, vascular dementia, dementia with Lewy bodies, frontotemporal dementia, or dementia arising from other diseases or conditions such as Parkinson's disease, vitamin B12 deficiency, thyroid abnormalities)
* Current residence in a skilled nursing facility
* Contraindication to undergoing MRI (eg, pacemaker [with the exception of an MRI-compatible pacemaker], severe claustrophobia, ferromagnetic implants such as a metal plate)
* Clinically significant congestive heart failure (eg, New York Heart Association [NYHA] Class III/IV symptoms or untreated Class II)
* Current atrial fibrillation of unstable angina (angina at rest) or history of myocardial infarction within the 12 months prior to screening
* Uncontrolled hypertension defined as systolic blood pressure > 160 mm Hg and/or diastolic > 100 mm Hg confirmed upon repeated measures
* History of thrombosis and/or thromboembolic disease (central or peripheral) within the 12 months prior to screening
* Known history of procoagulant abnormalities (eg, factor V Leiden, antiphospholipid syndrome, protein S/protein C deficiency, AT III deficiency)
* History of intracerebral hemorrhage within the 5 years prior to screening
* Evidence on MRI of: greater than 4 microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis, vasogenic edema, a macrohemorrhage, major stroke, prominent white matter disease with a rating score of 3 on the age-related white matter changes (ARWMC) scale from the European Task Force on ARWMC, or multiple lacunae (defined as more than 2 lacunae that are greater than 0.5 mm in size)
* Head trauma with loss of consciousness, contusion, or open head injury within the 12 months prior to screening
* Uncontrolled seizure disorder as defined by two or more breakthrough seizures per year despite adequate antiepileptic drug (AED) treatment
* Modified Hachinski score > 4 at time of screening
* Subjects with active malignancy or history of malignancy within 5 years prior to screening with the exception of the following: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment
* Active autoimmune or neuro-immunologic disorder
* Uncontrolled major depression, psychosis, or other major psychiatric disorder(s)
* Poorly controlled diabetes, defined as glycosylated (or glycated) hemoglobin (HbA1c) ≥ 6.5% at screening
* Creatinine clearance < 50% of normal adjusted for age and gender, as calculated according to the Cockcroft-Gault formula, at the time of screening
* Known history of untreated vitamin B12 deficiency within 6 months prior to screening, or clinically significant abnormally low vitamin B12 at the time of screening
* Abnormal clinical chemistry panel or hematology panel meeting any one of the following criteria:
* Serum alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN)
* Clinically significant anemia that precludes repeated blood sampling or hemoglobin (Hgb) < 10.0 g/dL
* Absolute neutrophil count (ANC) < 1000 cells/µL
* Known coagulopathy or platelet counts < 100,000 cells/µL
* Total serum protein > 9 g/dL
* Known history of or positive serology at screening for one or more of the following: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) type 1/2 antibody
* Immunoglobulin A (IgA) deficiency (< 8 mg/dL)
* Known history of hypersensitivity following infusions of human blood or blood components (e.g. human immunoglobulins or human albumin)
* Currently receiving or has received: anti-CD20 therapy within 12 months prior to screening, or other immunomodulatory therapies (e.g. anti-TNF, anti-IL-1, interferon) within 12 weeks prior to screening. The following exceptions are allowed: non-systemic corticosteroids (eg, topical, opthalmic or inhaled glucocorticoids) and low-dose systemic corticosteroids (prednisone < 10 mg/day or its equivalent)
* Currently receiving or has received intravenous or subcutaneous immunoglobulin treatment within the 2 years prior to screening, or has received immunoglobulin in Baxter Protocol 160701
* Currently receiving or has received at any time active immunization aimed at modulating AD progression
* Currently receiving or has received within 12 months prior to screening any investigational device, drug or biologic (eg passive immunotherapies with monoclonal or polyclonal antibodies) aimed at modulating AD progression
* Subject has been exposed to an investigational product (IP) or investigational device within 12 weeks prior to screening or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
* Subject is a family member or employee of the investigator
* The subject is nursing or intends to begin nursing during the course of the study
* Any disorder or disease, or clinically significant abnormality on laboratory or other clinical test(s) (eg, blood tests, urine tests, electrocardiogram, chest x-ray), that in medical judgment may impede the subject's participation in the study, pose increased risk to the subject, or confound the results of the study
* Currently receiving anti-coagulant agent and/or anti-platelet agent other than acetylsalicylic acid (a.k.a. aspirin)

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2012-01-23 (Actual); Primary Completion 2013-07-16 (Actual); Study Completion 2013-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (69):
- United States (37):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Long Beach, California
  - San Diego, California
  - Santa Ana, California
  - Boca Raton, Florida
  - Delray Beach, Florida
  - Edgewater, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Paducah, Kentucky
  - Saint Paul, Minnesota
  - Olive Branch, Mississippi
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Chester, New Jersey
  - Eatontown, New Jersey
  - Summit, New Jersey
  - Toms River, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Latham, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Providence, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Milwaukee, Wisconsin
- Woodville South, South Australia, Australia
- Belgium (5):
  - Edegem
  - Ghent
  - Hasselt
  - Leuven
  - Roeselare
- Canada (3):
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Sherbrooke, Quebec
- Japan (11):
  - Akashi
  - Akita
  - Azumino
  - Chiba
  - Fukui
  - Kyoto
  - Niigata
  - Osaka
  - Saga
  - Tokushima
  - Tokyo
- Poland (3):
  - Lublin
  - Ścinawa
  - Warsaw
- Spain (4):
  - Barakaldo, Vizcaya
  - Barcelona
  - Madrid
  - Valencia
- United Kingdom (5):
  - Uckfield, East Sussex
  - Bath
  - Brentford
  - Brighton
  - Glasgow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 58 clinical sites worldwide.
Pre-assignment Details: Of 508 enrolled subjects, 303 met entry criteria. 42 subjects discontinued before randomization due to study termination. Of 261 randomized subjects, 10 subjects discontinued before receiving treatment (7 study termination, 2 withdrawal by subject, 1 withdrawal by caregiver). Number of subjects who received treatment (IVIG,10% or placebo) = 251.
Period: Overall Study
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Started | 85 | 90 | 86
Received Treatment | 83 | 85 | 83
Completed | 0 (No subject completed the study as Baxter Healthcare terminated the study early.) | 0 (No subject completed the study as Baxter Healthcare terminated the study early.) | 0 (No subject completed the study as Baxter Healthcare terminated the study early.)
Not Completed | 85 | 90 | 86
Not completed — Withdrawal by Subject | 6 | 2 | 3
Not completed — Adverse Event | 5 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Study termination | 73 | 87 | 79
Not completed — Withdrawal by Caregiver | 0 | 0 | 2
Not completed — Use of prohibited medication | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises treated subjects (=safety analysis set).
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control | Total
Number analyzed (Participants) | 83 | 85 | 83 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (8.36) | 69.9 (8.59) | 70.6 (9.98) | 70.8 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 52 | 132
  Male | 40 | 48 | 31 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 1 | 3 | 1 | 5
  White | 81 | 79 | 78 | 238
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 67 | 66 | 199
  Canada | 8 | 7 | 7 | 22
  Spain | 3 | 5 | 3 | 11
  Belgium | 6 | 5 | 6 | 17
  Japan | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 18 in Cognitive Subscale of the Alzheimer´s Disease Assessment Scale (ADAS-Cog)
Description: The ADAS-Cog is a validated psychometric instrument that evaluates memory (word recall, word recognition), attention, reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). This test was administered by experienced raters certified by Alzheimer's Disease Cooperative Study (ADCS) at each site. Scores on the ADAS-Cog range from 0-70 with higher scores indicating greater impairment; hence increases from baseline reflect potential cognitive deterioration.
Time Frame: Baseline to 9 Months (actual time frame)
Population: Because this study was terminated early, 9-month analyses were conducted in the subset of participants that completed at least 9 months of treatment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 21 | 28 | 36
Scores on a scale | 4.0 (6.44) | 4.4 (8.56) | 3.1 (4.28)
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.243, Mixed Models Analysis; Difference in least square means = 1.4, 95% CI [-1.0 to 3.9]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.370, Mixed Models Analysis; Difference in least square means = 1.0, 95% CI [-1.2 to 3.3]

2. Primary Outcome: Change From Baseline to Month 18 in Alzheimer´s Disease Cooperative Study (ADCS)-Activities of Daily Living (ADL) Inventory
Description: The ADCS-ADL scale is a validated tool to assess instrumental and basic activities of daily living based on a 23 item structured interview of the caregiver or qualified study partner. Scores on the ADCS-ADL range from 0-78 with lower scores indicating greater impairment; hence decreases from baseline reflect potential functional deterioration.
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 21 | 29 | 36
Scores on a scale | -8.1 (7.36) | -5.0 (11.64) | -3.8 (9.26)
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis; Difference in least square means = -3.9, 95% CI [-7.4 to -0.3]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.586, Mixed Models Analysis; Difference in least square means = -0.9, 95% CI [-4.2 to 2.4]

3. Secondary Outcome: ADCS-Clinical Global Impression of Change (CGIC) at 18 Months
Description: The ADCS-CGIC is a validated categorical measure of change in a participant's global clinical status between baseline and follow-up visits, based on interview of the participant and the caregiver by a skilled and experienced clinician who was blinded to treatment assignment. The ADCS-CGIC score is based on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening).
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 10 | 16 | 16
Scores on a scale | 4.3 [3.7 to 4.8] | 4.4 [4.0 to 4.9] | 4.5 [4.1 to 5.0]
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.501, Mixed Models Analysis; Difference in least square means = -0.2, 95% CI [-1.0 to 0.5]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.783, Mixed Models Analysis; Difference in least square means = -0.1, 95% CI [-0.7 to 0.5]

4. Secondary Outcome: Change From Baseline to Month 18 in Neuropsychiatric Inventory (NPI)
Description: The NPI is a validated instrument used to assess behavioral psychopathology in AD; it evaluates the frequency and severity of 10 neuropsychiatric features including delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, sleep and night-time behavior change, and appetite and eating change. The NPI total score ranged 0-144, with higher scores indicating greater impairment.
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 21 | 29 | 36
Scores on a scale | 2.3 (5.76) | 3.8 (12.44) | 0.6 (5.68)
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis; Difference in least square means = 1.1, 95% CI [-2.6 to 4.7]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis; Difference in least square means = 3.7, 95% CI [0.3 to 7.1]

5. Secondary Outcome: Change From Baseline to Month 18 in Volumetric Magnetic Resonance Imaging (MRI) Parameters: Rate of Whole Brain Atrophy and Ventricular Enlargement
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 9 | 15 | 17
mm^3 | 0.00065 (0.00059) | 0.00057 (0.00070) | 0.00067 (0.00163)
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.593, ANCOVA; Difference in least square means = -0.00026, 95% CI [-0.00126 to 0.00073]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.940, ANCOVA; Difference in least square means = 0.00003, 95% CI [-0.00080 to 0.00086]

6. Secondary Outcome: Change From Baseline to Month 18 in Logsdon Quality of Life in Alzheimer´s Disease (QOL-AD)
Description: The QOL AD is a validated, 13-item instrument developed specifically for individuals with dementia. The assessment rates the participant´s quality of life for physical, emotional, interpersonal, and environmental domains. The QOL-AD total score ranged 13-52, with lower scores associated with a lower quality of life.
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 16 | 26 | 30
Scores on a scale | -0.1 (4.43) | 0.4 (3.68) | 0.1 (4.56)
Statistical Analysis 1: Comparison: IGIV, 10% at High Dose (0.4 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.633, Mixed Models Analysis; Difference in least square means = -0.5, 95% CI [-2.8 to 1.7]
Statistical Analysis 2: Comparison: IGIV, 10% at Low Dose (0.2 g/kg) vs Placebo Control; Test type: Superiority or Other; p = 0.981, Mixed Models Analysis; Difference in least square means = -0.0, 95% CI [-2.0 to 2.0]

7. Secondary Outcome: Change From Baseline to Month 18 in Impact of Alzheimer´s Disease on Caregiver Questionnaire (IADCQ)
Description: The IADCQ is a 12-item validated questionnaire that has been developed to measure the emotional, physical, and social impact of care giving on AD caregivers. Higher scores on the IADCQ are associated with a higher impact. IADCQ total score range: 0 (no impact) - 48 (greatest impact). Each item can be scored either 0 (Not at all), 1 (A little), 2 (Somewhat), 3 (A lot), or 4 (Extremely). As this is a 12-item scale, the minimum possible score is 0 and the maximum possible score is 4x12 = 48.
Time Frame: Baseline to 9 Months (actual time frame)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 19 | 27 | 30
Scores on a scale | 5.8 (4.13) | 1.9 (6.66) | 1.4 (5.97)

8. Secondary Outcome: Number of Participants Experiencing Study Product-related Adverse Events (AEs) and/or Serious Adverse Events (SAEs)
Time Frame: Throughout the study period: 18 Months
Population: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product.
Measure: Number; unit: participants
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
participants
  Participants with product-related AEs (incl SAEs) | 31 | 25 | 16
  Participants with product-related non-serious AEs | 30 | 25 | 16
  Participants with product-related SAEs | 1 | 0 | 1

9. Secondary Outcome: Number of Participants Experiencing Any AEs and/or SAEs
Time Frame: Throughout the study period: 18 Months
Population: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product.
Measure: Number; unit: participants
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
participants
  Participants with AEs (incl SAEs) | 57 | 54 | 49
  Participants with non-serious AEs | 55 | 53 | 48
  Participants with serious AEs (SAEs) | 5 | 7 | 7

10. Secondary Outcome: Number of Infusions Temporally Associated With AEs and/or SAEs
Description: A temporal association was defined as an AE and/or SAE occurring during or within 72 hours of completion of an infusion, regardless of causality.
Time Frame: During or within 72 hours of completion of an infusion
Population: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product.
Measure: Number; unit: infusions
Units Other Than Participants: Total number of infusions administered
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
Number analyzed (Total number of infusions administered) | 817 | 935 | 1023
infusions | 72 | 80 | 47

11. Secondary Outcome: Number of Infusions Associated With AEs and/or SAEs Occurring During or Within 7 Days of Completion of an Infusion
Time Frame: During or within 7 days of completion of an infusion
Measure: Number; unit: infusions
Units Other Than Participants: Total number of infusions administered
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
Number analyzed (Total number of infusions administered) | 817 | 935 | 1023
infusions | 97 | 107 | 72

12. Secondary Outcome: Number of Infusions Causally Associated With AEs and/or SAEs
Time Frame: Throughout the study period: 18 Months
Population: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product.
Measure: Number; unit: infusions
Units Other Than Participants: Total number of infusions administered
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
Number analyzed (Total number of infusions administered) | 817 | 935 | 1023
infusions | 46 | 48 | 30

13. Secondary Outcome: Number of Infusions Discontinued, Slowed, or Interrupted Due to an AE
Time Frame: Throughout infusions, approximately 2-5 hours
Population: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product.
Measure: Number; unit: infusions
Units Other Than Participants: Total number of infusions administered
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Number analyzed (Participants) | 83 | 85 | 83
Number analyzed (Total number of infusions administered) | 817 | 935 | 1023
infusions | 7 | 2 | 1

ADVERSE EVENTS:
Time Frame: Throughout the study period. The study was terminated early and no subject completed 18 months of treatment as planned per protocol. The duration of exposure to the investigational product varied for each subject.
Description: The safety analysis population includes the 251 subjects who received at least 1 infusion of investigational product (High Dose group: 83, Low Dose group: 85, Placebo group: 83).
Arm/Group | IGIV, 10% at High Dose (0.4 g/kg) | IGIV, 10% at Low Dose (0.2 g/kg) | Placebo Control
Serious Adverse Events (participants affected / at risk) | 5/83 | 7/85 | 7/83
Other Adverse Events (participants affected / at risk) | 30/83 | 33/85 | 30/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% at High Dose (0.4 g/kg) (N=83) | IGIV, 10% at Low Dose (0.2 g/kg) (N=85) | Placebo Control (N=83)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Human Ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus Ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV, 10% at High Dose (0.4 g/kg) (N=83) | IGIV, 10% at Low Dose (0.2 g/kg) (N=85) | Placebo Control (N=83)
Headache (Nervous system disorders) | 10 (14) | 11 (19) | 5 (6)
Fatigue (General disorders) | 5 (11) | 10 (15) | 6 (12)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 8 (9) | 1 (1)
Infusion Site Extravasation (General disorders) | 5 (10) | 6 (6) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (7) | 5 (7) | 3 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (4) | 5 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 10 (15)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 5 (5)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary and secondary outcome measures were originally planned to be assessed at 18 months. However, as the study was terminated early, an analysis was completed at 9 months instead, in a subset of subjects who had received 9 months of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, PIs are restricted from independently publishing results before completion of a single multicenter publication or one year after study completion, whichever occurs first. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (eg, for intellectual property protection).